CLINICAL TRIAL: NCT02611518
Title: A Phase 1, 2-Panel, Open-Label, Fixed-Sequence Study in Healthy Adult Subjects to Investigate the Pharmacokinetic Interaction Between JNJ-54861911 and Transporter Substrates Rosuvastatin and Metformin
Brief Title: A Pharmacokinetic Interaction Study Between JNJ-54861911 and Transporter Substrates Rosuvastatin and Metformin in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108091; 54861911ALZ1012 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2015-11-19; First posted 2015-11-20 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: Healthy; JNJ-54861911; Rosuvastatin; Metformin
MeSH Terms: interventions — Rosuvastatin Calcium; atabecestat; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- Panel 1 (Experimental): Participant will be administered a single oral dose of rosuvastatin 10 milligram (mg) on Day 1 and Day 14 and JNJ-54861911 at a dose of 25 mg once daily from Day 8 until Day 17.
  Interventions: Drug: Rosuvastatin; Drug: JNJ-54861911
- Panel 2 (Experimental): Participant will be administered a single oral dose of metformin 500-mg on Day 1 and Day 14 and JNJ-54861911 at a dose of 25 mg once daily from Day 8 until Day 16.
  Interventions: Drug: JNJ-54861911; Drug: Metformin

INTERVENTIONS:
Drug: Rosuvastatin — Rosuvastatin will be administered as a single oral 10 milligram (mg) dose on Day 1 and Day 14.
  Arms: Panel 1
Drug: JNJ-54861911 — JNJ-54861911 will be administered at a dose of 25 mg once daily from Day 8 to Day 17 (in panel 1), Day 8 to 16 (in panel 2).
Drug: Metformin — Metformin will be administered as a single oral 500 mg on Day 1 and Day 14.
  Arms: Panel 2

SUMMARY:
The purpose of this study is to look at how taking JNJ-54861911 every day will effect the amount of rosuvastatin or metformin in your blood after taking only a single dose of either one.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), single-center, fixed sequence, 2-panel study in a total of 32 healthy adult participants (16 participants per panel). The study consists of 3 phases: a Screening Phase of approximately 3 weeks (Days -22 to -2), an Open-Label Treatment Phase consisting of a single 19 day Treatment Period for Panel 1 (Days -1 to 18) or a single 18 day Treatment Period for Panel 2 (Days -1 to 17) and a Follow-up Phase of 5 to 7 days. In Panel 1, each participant will be administered a single oral dose of 10 milligram (mg) rosuvastatin on Day 1 and Day 14. Participants will receive JNJ-54861911 at a dose of 25 mg once daily from Day 8 until Day 17. In Panel 2, each participant will be administered a single oral dose of 500 mg metformin on Day 1 and Day 14. Participants will receive JNJ-54861911 at a dose of 25 mg once daily from Day 8 until Day 16. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Signed an informed consent document indicating they understand the purpose of and procedures required for the study and are willing to participate in the study
* Willing to adhere to the prohibitions and restrictions specified in this protocol
* All woman must have a negative serum pregnancy test at Screening and on Day minus (-) 1 of the Treatment Period
* If a woman must not be of childbearing potential: postmenopausal (greater than [>]45 years of age with amenorrhea for at least 12 months, or any age with amenorrhea for at least 6 months and a serum follicle stimulating hormone {FSH} level >40 International Units /Litre [IU/L]); documented permanently sterilized (example, tubal occlusion, hysterectomy, bilateral salpingectomy); or otherwise be incapable of pregnancy
* If a woman, must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for 3 months after receiving the last dose of study drug
* Non-smoker

Exclusion Criteria:

* Known allergy to rosuvastatin, metformin, JNJ-54861911 or to heparin or history of heparin induced thrombocytopenia
* History of or current clinically significant medical illness or a clinically significant 12-lead electrocardiogram (ECG) abnormality
* Donated blood or blood products or had substantial loss of blood (more than 500 milliliter [mL]) within 3 months before the first administration of study drug or intention to donate blood or blood products during the study
* Received an experimental drug or used an experimental medical device within 1 month or within a period less than 10 times the drug's half-life, whichever is longer, before the first dose of the study drug is scheduled
* Unable to swallow solid, oral dosage forms whole with the aid of water
* If a man, who plans to father a child while enrolled in the study or for 3 months after receiving the last dose of study drug
* Vulnerable participants
* Participants should not be enrolled if they have exposure to radiologic or magnetic resonance studies involving the use of intravascular contrast materials (for example, computed tomography [CT] scans with intravascular contrast materials), within 48 hours prior to Screening and for duration of study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2016-04-05 (Actual); Primary Completion 2016-06-14 (Actual); Study Completion 2016-06-14 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Up to Day 17
  The Cmax is the maximum observed concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Time (AUC [0-last]) | Up to Day 17
  The AUC (0-last) is the area under the plasma concentration-time curve from time zero to last quantifiable time.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) | Up to Day 17
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC (last) and C(last)/lambda(z); wherein AUC (last) is area under the plasma concentration time curve from time zero to last quantifiable time, C (last) is the last observed quantifiable concentration, and lambda (z) is elimination rate constant.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | Up to follow-up (5-7 Days after last dose of study drug administration)
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Berlin, Germany